CLINICAL TRIAL: NCT00537498
Title: Phase II Study of Urokinase Therapy for Treatment of Angiopathic or Angioneuropathic Diabetic Foot Syndrome
Brief Title: Urokinase Therapy in Diabetic Foot Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC-UK.2/AVK
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2007-09

CONDITIONS: Diabetic Foot; Arterial Occlusive Disease; Ischemia
Keywords: urokinase, diabetes, wound healing, major amputation
MeSH Terms: conditions — Diabetic Foot; Arterial Occlusive Diseases; Ischemia; Diabetes Mellitus | interventions — Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Interventional group
  Interventions: Drug: Urokinase

INTERVENTIONS:
Drug: Urokinase — Daily intravenous application of urokinase over 30 minutes
  Dosage:
  If plasma fibrinogen is > 2,5g/l application of 1 000 000 IU Urokinase If plasma fibrinogen is < 2,5g/l application of 500 000 IU Urokinase If plasma fibrinogen is < 1,6g/l treatment must be stopped and continued after rising up to >2g/l

SUMMARY:
The purpose of this study is to evaluate whether a treatment with urokinase (500 000 or 1 000 000 IU) can lead to ulcer-healing, lower rate of major amputation, and prolonged survival in patients with diabetic foot syndrome.

DETAILED DESCRIPTION:
Patients with diabetic foot ulceration and critical limb ischemia have a high risk of major amputation especially if limbs cannot be revascularized. Urokinase is effective in improving the microcirculation in critical limb ischemia by lowering fibrinogen and might improve outcomes. There are however no data on the efficacy and safety of urokinase treatment in terms of survival free of major amputation, ulcer healing and the rate of minor and major bleeding. Therefore this trial is conducted to investigate the effect of urokinase treatment on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* angiopathic or angioneuropathic diabetic foot lesions
* critical limb ischemia
* no surgical or interventional treatment option

Exclusion Criteria:

* feasibility of vascular surgery or angioplasty
* prior treatment of the current ulceration with urokinase
* need for dialysis
* creatinine > 180µmol/l
* any kind of cerebral event less than three months before inclusion into the study
* proliferative retinopathy (not remediated)
* uncontrolled hypertension
* hemorrhagic diathesis
* gastrointestinal bleeding
* need for oral anticoagulation
* mental disorders
* pregnancy
* participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2002-02; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of patients being alive, having no major amputation and healed ulceration | 12 months

SECONDARY OUTCOMES:
Each of overall survival, major amputation rate, survival free of major amputation rate, rate of ulcer healing, and safety | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian M. Schellong, Professor, Principal Investigator — Universitätsklinikum Carl Gustav Carus TU Dresden UniversitätsGefäßcentrum
Locations (1):
- Universitätsklinikum Carl Gustav Carus UniversitätsGefäßcentrum, Dresden, Germany